CLINICAL TRIAL: NCT00413140
Title: Biomarkers in Exhaled Breath Indicate Presence, Control and Severity of Cystic Fibrosis
Brief Title: Non-Invasive Biomarkers in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: AstraZeneca (Industry); Cystic Fibrosis Foundation (Other)
Other Study IDs: MEC 03-228-CF
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2006-12-19 (Estimated); Status verified 2003-11

CONDITIONS: Cystic Fibrosis
Keywords: childhood disease; cystic fibrosis; exhaled breath condensate; exhaled nitric oxide; airway inflammation; non-invasive inflammatory markers; controls; children
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background Chronic airway inflammation is present in cystic fibrosis. Non-invasive inflammometry may be useful in disease management.

Objective We studied 1) the ability of fractional exhaled nitric oxide and inflammatory markers (acidity, nitrite, nitrate, hydrogen peroxide, 8-isoprostane, interferon-γ, tumor necrosis factor-α, interleukin-2,-4,-5,-10) in exhaled breath condensate, to discriminate between cystic fibrosis and control children, and, 2) the relationship of biomarkers with control and severity of cystic fibrosis.

Methods In 98 children (48 cystic fibrosis / 50 controls), condensate was collected using a glass condenser. Exhaled nitric oxide was measured using the NIOX®.

ELIGIBILITY:
Inclusion Criteria:

CF population

* Children known with CF were recruited from the outpatient clinics. CF disease was defined as a combination of typical clinical features (e.g. persistent pulmonary problems, meconium ileus, failure to thrive, steatorrhoe) and an abnormal sweat test (Chloride > 60 mM). Uncontrolled CF was diagnosed by the paediatric pulmonologist based on a change in the presence or severity of respiratory symptoms in association with CF, and/or a decrease in lung function parameters compared to previous measurements during the last four weeks.

Control population

* Control children without lung disease were recruited from the outpatient clinic of the University Hospital Maastricht. The reasons of consultation were constipation and enuresis nocturna. All children completed the 'International Study of Asthma and Allergies in Childhood (ISAAC) questionnaire to exclude children with any (history of) airway or allergy complaints, in order to exclude asthmatic disease

Exclusion Criteria:

For both study populations:

* Diseases that may interfere with the results of the study (e.g. upper airway infection, heart disease, anatomic abnormalities of the airways and other chronic inflammatory diseases, such as Crohns disease and rheumatoid arthritis)
* Mental retardation
* Inability to perform the EBC collection procedure
* Active smoking
* Use of the following medication: papaverin, sodium nitroprusside, angiotensin-converting enzyme (ACE) inhibitors, oxymetazoline, L-arginine, or nitric oxide synthase (NOS) inhibitors.

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 2004-06; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte M Robroeks, M, Principal Investigator — Maastricht University Medical Center; Edward Dompeling, MD, PhD, Study Director — Maastricht University Medical Center; Quirijn Jöbsis, MD, PhD, Study Director — Maastricht University Medical Center
Locations (4):
- Netherlands (4):
  - Catharina Hospital, Eindhoven
  - University Hospital Maastricht, Maastricht
  - St Radboud Childrens Hospital, Nijmegen
  - Máxima Medical Centre, Veldhoven